CLINICAL TRIAL: NCT02530112
Title: Functional Outcome Measures for Head and Neck Patients
Status: Terminated | Type: Observational
Why Stopped: The study proved very difficult to do on paper surveys. The health system is now doing these via the chart with more success.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 17913
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2023-08

CONDITIONS: Otorhinolaryngology Subjects Undergoing Free Flap Surgery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Phase 1: First round of survey respondents.
  Interventions: Other: Survey
- Phase 2: Second round of survey respondents.
  Interventions: Other: Survey
- Phase 3: Third round of survey respondents.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
The objective of this study is to identify outcome measures for cancer control in Head and Neck cancer patient populations at the University of Pennsylvania (HUP, PAH, Presby) by administering various functional outcome surveys and questionnaires about their reconstructive surgery. We hope to ultimately develop a QOL indicator that will reflect the impact of reconstructive surgery on patient's quality of life, and help with therapeutic interventions and explanation of expectations prior to surgery.

DETAILED DESCRIPTION:
Few studies examine quality of life outcome measures with initial diagnosis, surgical procedures,perioperative measures (such as use of perioperative blood transfusion or pressors), and outcomes for cancer control and free flap survival. This sub-protocol, in conjunction with protocol #816676 (Otorhinolaryngology Research Registry) will serve as a hypothesis generating study for future research on reconstructive free flap surgery outcomes by narrowing down existing questionnaires to tailor it specifically for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have consented to Otorhinolaryngology Research Registry and are undergoing free flap surgery.

Exclusion Criteria:

* No children, pregnant women, or prisoners will be consented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have consented to Otorhinolaryngology Research Registry and are undergoing free flap surgery.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-02-02 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Completion of Survey | 9 years
  Completion of quality of life surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cannady, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States